CLINICAL TRIAL: NCT03574883
Title: Effects of the Transcranial Alternative Electric Stimulation on the Consciousness Access in Healthy Subjects
Brief Title: Consciousness Transcranial Alternative Electric STimulation
Acronym: CONTEST_1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: C17-22; 2017-A02761-52 (Registry Identifier: IDRCB)
Record Dates: First submitted 2018-04-19; First posted 2018-07-02 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Conscious access; transcranial electric stimulation; tACS; Global neuronal workspace; Masking paradigm; tDCS
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This study is composed of two independent sub-studies, one exploring the effects of tACS and the other the effects of tDCS, with different participants assigned to the two sub-studies. There will be 3 arms in tACS group and 2 arms in tDCS group. Among each sub-study, all participants will participate in all arms (hence the cross-over design).
Who Masked: Participant, Investigator
Masking Description: Study will be double-blind : neither participant nor the investigator will know which stimulation type (in-phase active, anti-phase active or sham) is on.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- In-phase tACS (Experimental): 6 Hz stimulation (1000 μA) will be applied simultaneously over the left prefrontal dorso-lateral cortex (F3 of the 10-20 international scalp EEG system) and the left parietal cortex (P3) for 20 minutes using an 8-channels stimulator. The phase difference between the two stimulation sites will be 0°.
  Interventions: Device: tACS
- Anti-phase tACS (Active Comparator): 6 Hz stimulation (1000 μA) will be applied simultaneously over the left prefrontal dorso-lateral cortex (F3 of the 10-20 international scalp EEG system) and the left parietal cortex (P3) for 20 minutes using an 8-channels stimulator. The phase difference will be 180°,
  Interventions: Device: tACS
- Sham tACS (Sham Comparator): The stimulation (anti-phase) will start with a current intensity of 1000 μA lasting for 30 seconds. Afterwards, the intensity will progressively decrease over 20 seconds until cessation.
  Interventions: Device: tACS
- Active tDCS (Experimental): 1000 μA tDCS stimulation will be applied simultaneously over the left prefrontal dorso-lateral cortex (F3 of the 10-20 international scalp EEG system) and the left parietal cortex (P3) for 20 minutes using an 8-channels stimulator
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): The stimulation will start with a current intensity of 1000 μA lasting for 30 seconds. Afterwards, the intensity will progressively decrease over 20 seconds until cessation.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tACS — tACS is a non-invasive stimulation technique that works by delivering a weak sinusoidally oscillating electrical current to the surface of the skull to entrain oscillations in the brain.
  Arms: Anti-phase tACS; In-phase tACS; Sham tACS
Device: tDCS — tDCS is a form of neuromodulation method where very low levels of constant current are delivered to specifically targeted areas of the brain
  Arms: Active tDCS; Sham tDCS

SUMMARY:
The aim of this study is to investigate the effect of transcranial Alternating Current Stimulation (tACS) at theta frequency and the the effect of transcranial Direct Current Stimulation (tDCS) on the conscious access to visual stimuli. tACS and tDCS are non-invasive stimulation techniques that are used to induce brain oscillations at certain frequency or to increase the brain activity in applied region. Healthy participants will perform a behavioral task measuring conscious access (visual backward metacontrast masking task) before, during and after fronto-parietal tACS or tDCS stimulation which will increase neural activity in the two sites. This will allow us to examine online and remaining effects of the stimulation and the causal role of fronto-parietal activity on conscious access.

DETAILED DESCRIPTION:
Behavioral task

The behavioral task consists in presentation of a para-foveal numerical target on a screen for 16 ms either right or left of a central fixation point, followed by a visual mask, made of letters surrounding the target, presented for 250 ms. The delay between the target and the mask (Stimulus Onset Asynchrony - SOA) will be variable (16 ms, 33 ms, 50 ms, 66 ms or 83 ms). Participants will then be asked to perform two tasks. First (objective task), participants will be asked to indicate as quickly as possible whether the target was bigger or smaller than the digit "5". Second (subjective task), they will be requested to judge the visibility of the presented target by indicating whether they had seen the target or not.

tACS

Study design

The study design is composed of three experimental sessions. In these sessions, participants will first complete the behavioral paradigm as presented above while having their brain activity recorded with EEG. Afterwards, they will re-perform the task during and after tACS stimulation. tACS stimulation type will differ in each session : in-phase, anti-phase or sham (see below for further details). Stimulation sessions will occur in a double-blind randomized crossover design (neither the participant nor the experimenter knows which session includes which stimulation type), with at least 2 days of interval between them.

Stimulation

During tACS sessions, 6 Hz stimulation (1000 μA) will be applied simultaneously over the left prefrontal dorso-lateral cortex (F3 of the 10-20 international scalp EEG system) and the left parietal cortex (P3) using an 8-channels stimulator (Starstim NE, Neuroelectrics, Barcelona, Spain) with small round sponge electrodes (25 cm2 surface, maximal current density of 0.06 μA/cm2), controlled via Bluetooth. In the in-phase condition, the phase difference between the two stimulation sites will be 0° which will entrain synchronization between sites. In the anti-phase condition on the other hand, the phase difference will be 180°, which should desynchronize the activity in the two cortices. In the sham condition, the stimulation (also anti-phase) will start with a current intensity of 2000 μA lasting for 30 seconds. Afterwards, the intensity will progressively decrease over 20 seconds until cessation. Each stimulation session will take 20 minutes and the positions of stimulation electrodes and the duration of the stimulation will be kept identical for all conditions.

tDCS

Study design

The study is composed of two experimental sessions: one tDCS session and one sham session. In the tDCS session, participants will do the behavioral task (with an EEG recording) during and after 20 minutes of 1000 μA tDCS stimulation. As a control, participants will do the behavioral task in a second session (sham session) during which they will have a sham stimulation instead of tDCS stimulation. The two sessions will occur in a double-blind randomized crossover design (neither the participant nor the experimenter knows which session includes which stimulation type), with at least 2 days of interval between them.

Stimulation

During tDCS session, 1000 μA stimulation will be applied simultaneously over the left prefrontal dorso-lateral cortex (F3 of the 10-20 international scalp EEG system) and the left parietal cortex (P3) using an 8-channels stimulator (Starstim NE, Neuroelectrics, Barcelona, Spain) with small round sponge electrodes (25 cm2 surface, maximal current density of 0.06 μA/cm2), controlled via Bluetooth. In the sham condition, the stimulation will start with a current intensity of 1000 μA lasting for 30 seconds. Afterwards, the intensity will progressively decrease over 20 seconds until cessation. The reason for this subtle manipulation is to make sure that participants will be unable to notice the difference between active tDCS and sham tDCS stimulation. Each stimulation session will take 20 minutes and the positions of stimulation electrodes and the duration of the stimulation will be kept identical for all conditions.

ELIGIBILITY:
Inclusion Criteria:

* French social security affiliation
* Absence of neurological and psychiatric disorders
* Absence of antiepileptic treatment
* Normal vision (with or without correction)
* Age between 18 and 60 years
* Right-handedness
* Signed informed consent to participate

Exclusion Criteria:

* Person under legal protection (legal guardian, tutor, curator)
* Past medical history of epilepsy
* Past medical history of neurological or psychiatric disorders
* Electrical stimulation contraindication (metallic intra-cranial implants, pacemaker or implantable cardioverter-defibrillator, cranial prosthesis)
* Antiepileptic and other psychotropes treatment
* Pregnant, parturient or breastfeeding women
* Left-handedness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2021-07-16 (Actual)

PRIMARY OUTCOMES:
Change in subjective performance on the behavioral task (% of seen masked target) between before and after stimulation. | Measured at each stimulation sessions (three sessions in a randomized cross-over order) for each participant. The three sessions will span in an average of two weeks.
  Change in the percentage of the correct responses on the subjective evaluation, that is the percentage of seen masked target at each SOA over all masked target presented, between before and after stimulation, for each stimulation modality (inphase theta, antiphase theta, sham).

SECONDARY OUTCOMES:
Change in visual evoked potentials between before and after stimulation. | Measured at each stimulation sessions (three sessions in a randomized cross-over order) for each participant. The three sessions will span in an average of two weeks.
  Change in amplitudes and delays of event related potentials evoked by the target at different SOA and according to the visibility (P1, N1, N2, P300) between before and after stimulation for each stimulation modality.
Change in quantitative EEG measures between before and after stimulation. | Measured at each stimulation sessions (three sessions in a randomized cross-over order) for each participant. The three sessions will span in an average of two weeks.
  Changes in quantitative EEG measures (spectral power, complexity, connectivity) between before and after stimulation for each stimulation modality.
Change in objective performance on the behavioral task (% of correct response on the number comparison task for masked target) between before and after stimulation. | Measured at each stimulation sessions (three sessions in a randomized cross-over order) for each participant. The three sessions will span in an average of two weeks.
  Change in the percentage of the correct responses on the objective comparison task, that is the percentage of correct response on the number comparison task for masked target at each SOA, between before and after stimulation, for each stimulation modality (inphase theta, antiphase theta, sham).

CONTACTS AND LOCATIONS:
Overall Officials: Lionel NACCACHE, MD, PhD, Principal Investigator — CR-ICM U 975 /UMRS INSERM 1127; Jacobo D SITT, MD, PhD, Principal Investigator — CR-ICM U 975 /UMRS INSERM 1127; Bertrand HERMANN, MD, Study Chair — CR-ICM U 975 /UMRS INSERM 1127
Locations (1):
- Institut du Cerveau et de la Moelle - CR-ICM U 975 / UMRS INSERM 1127, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Del Cul A, Baillet S, Dehaene S. Brain dynamics underlying the nonlinear threshold for access to consciousness. PLoS Biol. 2007 Oct;5(10):e260. doi: 10.1371/journal.pbio.0050260. PMID 17896866
- [Background] Polania R, Nitsche MA, Korman C, Batsikadze G, Paulus W. The importance of timing in segregated theta phase-coupling for cognitive performance. Curr Biol. 2012 Jul 24;22(14):1314-8. doi: 10.1016/j.cub.2012.05.021. Epub 2012 Jun 7. PMID 22683259